CLINICAL TRIAL: NCT01785199
Title: Effects of Head Elevation by an Adjustable Bed on Sleep-disordered Breathing
Brief Title: Effects of Head Elevation by a Bed on Sleep-disordered Breathing
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: Seda Chemical Products Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Ching-Lung Liu, MD, Mackay Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UWB-C-008
Record Dates: First submitted 2013-01-31; First posted 2013-02-07 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Sleep-disordered Breathing; Obstructive Sleep Apnea
Keywords: apnea-hypopnea index; obstructive sleep apnea; body posture; ultra-wideband
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- normal (AHI < 5) (Placebo Comparator): Patients who are eligible for this study will sleep on an automatic adjustable bed with a second PSG performed within the next one month.
  Interventions: Procedure: Head elevation by an automatic adjustable bed
- mild OSA (AHI between 5 and 15) (Active Comparator): Patients who are eligible for this study will sleep on an automatic adjustable bed with a second PSG performed within the next one month.
  Interventions: Procedure: Head elevation by an automatic adjustable bed
- moderate OSA (AHI between 15 and 30) (Active Comparator): Patients who are eligible for this study will sleep on an automatic adjustable bed with a second PSG performed within the next one month.
  Interventions: Procedure: Head elevation by an automatic adjustable bed
- severe OSA (AHI > 30) (Active Comparator): Patients who are eligible for this study will sleep on an automatic adjustable bed with a second PSG performed within the next one month.
  Interventions: Procedure: Head elevation by an automatic adjustable bed

INTERVENTIONS:
Procedure: Head elevation by an automatic adjustable bed — The automatic device is initiated when the patient suffers from apnea ≥ 10 seconds, which is detected by an ultra-wideband (UWB) sensor placed under the bed. The head will be slightly elevated at an angle of 10 degrees lasting 10 seconds and then be put down softly.

SUMMARY:
Sleep is known to be a dynamic state of consciousness that is characterized by rapid fluctuations in autonomic activity as well as changes in body postures. Body postures during sleep influence the severity of sleep-disordered breathing because a supine position is associated with an increase in upper airway collapsibility and thus an increase in frequency and duration of snoring and apnea. Use of an adjustable bed to elevate patients' head might improve those conditions. The purpose of the present study is to determine whether use of an automatic adjustable bed is associated with reducing sleep-disordered breathing in patients with suspected obstructive sleep apnea (OSA) due to upper airway problems.

DETAILED DESCRIPTION:
From the Chest and Otorhinolaryngology Department, patients with symptomatic sleep-disordered breathing will be referred to the Sleep Center. After an interview these subjects will undergo a full-night polysomnography (PSG). Patients who are eligible for this study will sleep on an automatic adjustable bed with a second PSG performed within the next one month. The automatic device is initiated when the patient suffers from apnea ≥ 10 seconds, which is detected by an ultra-wideband (UWB) sensor placed under the bed. The head will be slightly elevated at an angle of 10 degrees lasting 10 seconds and then be put down softly. Parameters of sleep efficiency and architecture, apnea-hypopnea index (AHI), and oxygen saturation will be obtained during each PSG. According to the severity, enrolled patients will be classified into 4 groups as normal (AHI < 5), mild OSA (AHI between 5 and 15), moderate OSA (AHI between 15 and 30) and severe OSA (AHI > 30).

Using an automatic adjustable bed will improve sleep-disordered breathing with a reduction of AHI score is assumed. The minimal sample size is estimated to be 14 subjects per group with the intention of providing 80% power and an overall two-sided 5% type I error. A total of 60 subjects (15 subjects per group) will be enrolled to achieve the necessary number of evaluable subjects, anticipating roughly a 10% drop-out rate.

Informed written consent will be obtained from all subjects. This study was approved by the Mackay Memorial Hospital Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

* Subjects known to have snoring or sleep-disordered breathing

Exclusion Criteria:

* Refusal to participate
* Pregnancy
* Psychiatric disorders
* Clinical instability in the previous month

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of AHI score. | Two full-night PSGs will be performed within one month
  Using an automatic adjustable bed will improve sleep-disordered breathing with a reduction of AHI score is assumed.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Lung Liu, MD, Principal Investigator — Sleep Center, Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Tamshui Branch, New Taipei City, Taiwan